CLINICAL TRIAL: NCT00810290
Title: Lawrence Latino Diabetes Prevention Project
Acronym: LLDPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Ira S. Ockene, M.D., University of Massachusetts Medical School
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: H-11214; DK67549
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Latino health; Community participatory research; Translational Research
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: lifestyle intervention — A group-based intervention including 13 group sessions complemented by three individual home visits was developed using principles of social learning theory and patient-centered counseling. The intervention was intended to increase awareness of diabetes prevention strategies, foster positive diabetes prevention attitudes (i.e., self-efficacy) and promote healthy lifestyle behaviors in the target Latino population using literacy-sensitive and culturally-tailored strategies and materials.

SUMMARY:
The Lawrence Latino Diabetes Prevention Project (LLDPP) is a community-based translational research study which aims to reduce the risk of diabetes among Latinos who have a >30% probability of developing diabetes in the next 7.5 years per a predictive equation. The project was conducted in Lawrence, Massachusetts; a predominantly Caribbean-origin urban Latino community. Individuals were identified primarily from a community health center's patient panel, screened for study eligibility, randomized to either a usual care or a lifestyle intervention condition, and followed for one year.

DETAILED DESCRIPTION:
The group format of the intervention included 13 group sessions complemented by 3 individual home contacts over one year and was implemented by individuals from the community with training and supervision by a clinical research nutritionist and a behavioral psychologist. Study measures included demographics, Stern predictive equation components (age, gender, ethnicity, fasting glucose, systolic blood pressure, HDL-cholesterol, body mass index, and family history of diabetes), glycosylated hemoglobin, dietary intake, physical activity, depressive symptoms, social support, and quality of life. Body weight was measured at baseline, 6-months, and one-year; all other measures were assessed at baseline and one-year. All surveys were orally administered in Spanish.

ELIGIBILITY:
Inclusion Criteria:

* Is Latino/Hispanic;
* Has a 7.5 year likelihood of becoming diabetic of greater than or equal to 30% as predicted by the Stern formula;
* Is greater than or equal to 25 years of age;
* Has a BMI greater than or equal to 24 kg m2.

Exclusion Criteria:

* An inability or unwillingness to give informed consent;
* Has clinically diagnosed diabetes, or a fasting blood sugar of greater than or equal to 126 mg/dl;
* Plans to move out of the area within the study period;
* Has a psychiatric illness which limits ability to participate;
* Has no telephone;
* Is unable to walk unaided, or cannot walk five city blocks (1/4 mile) without stopping;
* Is not cleared for the PA component by the pt's GLFHC primary care provider;
* Has a medical conditions likely to limit lifespan;
* Is on medications or has a medical condition that interfere with the assessment for diabetes.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2004-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Weight loss. | 1 year
HgbA1c | 1 year

SECONDARY OUTCOMES:
Change in fasting blood sugar. | 1 year
Changes in LDL- and HDL-cholesterol. | 1 year
Change in blood pressure. | 1 year
Change in depression. | 1 year
Change in quality of life. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ira S Ockene, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- Lawrence Senior Center, Lawrence, Massachusetts, United States

REFERENCES:
- [Background] Olendzki BC, Ma Y, Hebert JR, Pagoto SL, Merriam PA, Rosal MC, Ockene IS. Underreporting of energy intake and associated factors in a Latino population at risk of developing type 2 diabetes. J Am Diet Assoc. 2008 Jun;108(6):1003-8. doi: 10.1016/j.jada.2008.03.006. PMID 18502234
- [Derived] Ockene IS, Tellez TL, Rosal MC, Reed GW, Mordes J, Merriam PA, Olendzki BC, Handelman G, Nicolosi R, Ma Y. Outcomes of a Latino community-based intervention for the prevention of diabetes: the Lawrence Latino Diabetes Prevention Project. Am J Public Health. 2012 Feb;102(2):336-42. doi: 10.2105/AJPH.2011.300357. Epub 2011 Dec 15. PMID 22390448
- [Derived] Merriam PA, Tellez TL, Rosal MC, Olendzki BC, Ma Y, Pagoto SL, Ockene IS. Methodology of a diabetes prevention translational research project utilizing a community-academic partnership for implementation in an underserved Latino community. BMC Med Res Methodol. 2009 Mar 13;9:20. doi: 10.1186/1471-2288-9-20. PMID 19284663